CLINICAL TRIAL: NCT04950556
Title: The Effects of Pelvic Floor Muscle Training in Women With Overactive Bladdder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, associate professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/06/27
Record Dates: First submitted 2021-06-27; First posted 2021-07-06 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-06

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups (control and exercise) for treatment.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Fast and slow contractions will be taught in PFMT. For fast contractions, they will be asked to contract and relax the pelvic floor muscles quickly. For slow contractions, they will be asked to contract the pelvic floor muscles slowly, keep them at maximum contraction and relax slowly. Ten slow contractions in addition to 10 fast contractions will be considered as 1 set of exercises. For the first week, they will be asked to do 5 sets of exercises per day, every day. Then, the number of sets will be increased by 5 each week and the number of sets will reach 30 in the 6th week. PFMT will be applied by the patients as a home program every day of the week for 6 weeks.
  Interventions: Other: Exercise
- Control group (Other): Waiting list will included in control group.
  Interventions: Other: Control

INTERVENTIONS:
Other: Exercise — Pelvic floor muscle exercise will be given to the exercise group
  Arms: Exercise group
Other: Control — No intervention
  Arms: Control group

SUMMARY:
The aim of our study is to investigate the effects of pelvic floor muscle training (PFMT) on pelvic floor muscle strength, sexual functions, bladder symptoms and quality of life in women with overactive bladder (OAB).

DETAILED DESCRIPTION:
Overactive bladder (OAB) is defined by the International Continence Association as an "urgency with or without urge urinary incontinence, often accompanied by frequency and nocturia." Accordingly, pelvic floor muscle training (PFMT) plays an important role in the management of OAB. However, a recent systematic review suggests that PFMT is insufficient against OAB.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of overactive bladder
* Being volunteer

Exclusion Criteria:

* have a neurological disorder
* only those with stress urinary incontinence
* presence of advanced pelvic organ prolapse (stage 3-4)
* Having a mental problem that will prevent cooperation in evaluation and / or applications
* Women with the presence of malignant condition

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle strength | change from baseline at 6 weeks
  The pelvic floor muscle strength of the patients will be evaluated by digital palpation. Change in pelvic floor muscle strength as measured with the Modified Oxford Scale, which ranges from 0 to 5
Sexual Function | change from baseline at 6 weeks
  Female sexual function will be assessed using the Female Sexual Function Index. This 19-question questionnaire deals with the subject in a multidimensional way by questioning the states of desire, arousal, lubrication, orgasm, satisfaction and pain. The highest raw score that can be obtained from the questionnaire is 95, and the lowest raw score is 4.

SECONDARY OUTCOMES:
OAB symptoms | change from baseline at 6 weeks
  OAB symptoms will be evaluated OAB-V8. There are 8 questions in this form and the answers given to each question are scored between 0 and 5. The scores that can be obtained from the entire scale range from 0 to 40.
Urinary frequency, nocturia and the number of urinary incontinence | change from baseline at 6 weeks
  Patients will be also instructed to keep voiding diary
Life quality | change from baseline at 6 weeks
  Life quality will be assessed with King's Health Questionnaire (KHQ).This questionnaire consists of two parts and 32 items.. The minimum possible score is 0 (best health) and the maximum possible score is 100 (worst health).

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University